CLINICAL TRIAL: NCT06849362
Title: A Multicenter Retrospective Study on Optimizing Combination Immunotherapy Strategies for MSS/MSI-L/pMMR Advanced Colorectal Cancer: Comprehensive Clinical and Prognostic Analysis
Brief Title: Multicenter Retrospective Study on Optimizing Combination Immunotherapy Strategies in MSS/MSI-L/pMMR Advanced Colorectal Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Yue Gou (Other)
Responsible Party: Sponsor-Investigator, Yue Gou, MD, Central South University
Organization: Central South University (Other)
Other Study IDs: 20240306-MSS-Gou
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Colorectal Cancer (CRC); MSS Metastatic Colorectal Cancer; Immunotherapy
Keywords: MSS Colorectal Cancer; MSI-L Colorectal Cancer; pMMR Colorectal Cancer; Combination Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Immunotherapy + Bevacizumab Group: Immunotherapy + Bevacizumab Group
  Interventions: Drug: Bevacizumab
- Immunotherapy only Group: Immunotherapy only
- Immunotherapy + Chemotherapy + Bevacizumab Group: Immunotherapy + Chemotherapy + Bevacizumab
  Interventions: Drug: Bevacizumab
- Chemotherapy only Group: Chemotherapy only

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is an anti-vascular endothelial growth factor (VEGF) monoclonal antibody used in combination with chemotherapy or immunotherapy for the treatment of metastatic colorectal cancer (CRC). In this study, bevacizumab is administered as part of combination therapy in certain patient groups to assess its impact on treatment efficacy in MSS/MSI-L/pMMR advanced colorectal cancer.
  Patients receiving bevacizumab will be evaluated for treatment response, survival outcomes, and potential biomarkers predictive of therapeutic efficacy. The study will compare the clinical benefits of immunotherapy alone, immunotherapy + bevacizumab, and immunotherapy + chemotherapy + bevacizumab to determine the optimal treatment strategy.
  The dose and administration schedule of bevacizumab will follow standard clinical guidelines as per institutional protocols.
  Groups: Immunotherapy + Bevacizumab Group; Immunotherapy + Chemotherapy + Bevacizumab Group

SUMMARY:
This multicenter retrospective study aims to evaluate and optimize combination immunotherapy strategies for patients with microsatellite stable (MSS), microsatellite instability-low (MSI-L), or mismatch repair-proficient (pMMR) advanced colorectal cancer (CRC). The study will analyze clinical outcomes, treatment responses, and prognostic factors in patients who received various immunotherapy regimens. Data from multiple institutions will be collected to identify potential predictive biomarkers and effective therapeutic combinations. The findings may provide critical insights for improving immunotherapy strategies in MSS/MSI-L/pMMR CRC patients.

DETAILED DESCRIPTION:
This multicenter retrospective cohort study aims to evaluate the effectiveness of combination immunotherapy strategies in microsatellite stable (MSS), microsatellite instability-low (MSI-L), and mismatch repair-proficient (pMMR) advanced colorectal cancer (CRC) patients. Given the limited response of these CRC subtypes to immune checkpoint inhibitors (ICIs) alone, this study seeks to identify optimal combination regimens that can enhance therapeutic efficacy.

Study Objectives:

1. To assess clinical outcomes (e.g., overall survival, progression-free survival, objective response rate) in patients receiving different immunotherapy combinations.
2. To evaluate predictive biomarkers that may influence treatment response in MSS/MSI-L/pMMR CRC.
3. To compare the efficacy of various immunotherapy-based regimens, including ICIs combined with chemotherapy, targeted therapy, or anti-angiogenic agents like bevacizumab.

Methods:

* Data Source: Patient records from multiple institutions will be retrospectively analyzed.
* Patient Population: Individuals diagnosed with MSS/MSI-L/pMMR advanced CRC who have received at least one line of immunotherapy-based combination treatment.
* Data Collection: Demographics, tumor characteristics, treatment regimens, survival outcomes, and biomarker profiles.
* Statistical Analysis: Kaplan-Meier survival analysis, Cox proportional hazards model, and subgroup analyses based on biomarker expression.

Eligibility Criteria:

Approval was obtained from the institutional review boards of all four centers, adhering to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines and reported in accordance with the STROCSS 2024 criteria. Informed consent was not required.

* Inclusion Criteria:

  * Patients with MSS metastatic colorectal cancer who underwent immunotherapy.
  * Comprehensive collection of demographic and molecular characteristics.
  * Patients were included irrespective of treatment context.
* Exclusion Criteria:

  * Individuals lacking definitive pathological diagnosis.
  * Patients without response evaluation data.
  * Cases missing pertinent follow-up information.

Treatment Response Evaluation:

Treatment responses were evaluated radiographically according to the Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 guidelines.

Ethical Considerations:

Ethical approval was obtained from the institutional ethics committee of our hospital, ensuring compliance with ethical and regulatory standards for retrospective studies.

Expected Outcomes:

The study aims to identify effective treatment strategies for MSS/MSI-L/pMMR CRC patients, provide real-world evidence on the role of combination immunotherapy, and explore potential predictive biomarkers to improve patient selection for immunotherapy-based approaches.

This research will contribute to optimizing treatment strategies for immunotherapy-resistant CRC subtypes and guide future clinical trials.

ELIGIBILITY:
Inclusion Criteria:1) study subjects were mCRC patients with explicitly stated MSS/MSI-L/pMMR status; 2) at least one cohort included immunotherapy treatment; 3); primary outcomes of this study were defined as Disease Control Rate (DCR) and Progression-Free Survival (PFS); secondary outcomes included Objective Response Rate (ORR), Overall Survival (OS), and Adverse Drug Reactions (ADRs) Exclusion Criteria: individuals lacking definitive pathological diagnosis, response evaluation, or pertinent follow-up data

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes patients diagnosed with microsatellite stable (MSS), microsatellite instability-low (MSI-L), or mismatch repair-proficient (pMMR) metastatic colorectal cancer (CRC) who have undergone immunotherapy-based treatment. Eligible participants are those who received immune checkpoint inhibitors (ICIs) alone or in combination with chemotherapy and/or bevacizumab as part of their treatment regimen.
  Patients were enrolled from multiple medical centers, with data collected retrospectively. Inclusion criteria require a confirmed pathological diagnosis of MSS/MSI-L/pMMR CRC, available treatment and follow-up data, and a history of receiving at least one immunotherapy-based regimen. Exclusion criteria include patients lacking complete clinical records, follow-up data, or radiographic response assessments.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 02/28/2024
  Disease Control Rate (DCR)
Progression-Free Survival | 02/28/2024
  Progression-Free Survival (PFS)

SECONDARY OUTCOMES:
Objective Response Rate | 02/28/2024
  Objective Response Rate (ORR)
Overall Survival | 02/28/2024
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya hospital, CSU, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
Since the data collection and analysis for this study are ongoing, the decision on sharing individual participant data (IPD) has not been finalized. Data sharing will be considered in accordance with institutional policies, ethical guidelines, and patient confidentiality regulations. If data sharing is approved in the future, details regarding access and sharing mechanisms will be specified accordingly.